CLINICAL TRIAL: NCT05250362
Title: Non-feeder Cell ex Vivo Expanded Allogeneic NK Cells Infusion Decrease Relapse Post Hematopoietic Stem Cell Transplantation.
Brief Title: Ex Vivo Expanded NK Cells Infusion Decrease Relapse Post Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principal Investigator, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNKI1.0
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Hematologic Malignancy
Keywords: NK cell; stem cell transplant; relapse
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Intervention Model Description: intervention: Expanded NK cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — MYELOABLATIVE CONDITIONING REGIMEN: Patients with myeloid malignancies receive busulfan on days -7 to -4, fludarabine IV over 1 hour on days -7 to -3, cytarabine IV over 4 hours on days -7 to -3. Patients with lymphoproliferative disorders receive busulfan on day -7 to -4, cladribine IV over 1 hour on days -7 to -3, gemcitabine IV over 4 hours on days -7 and -3.
  TRANSPLANT: Patients undergo PBSC transplant on day 0.
  POST-TRANSPLANT CYCLOPHOSPHAMIDE AND GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days 3 and 4, cyclosporin IV beginning on day 5 for 2 weeks and then PO for approximately 4 months, and mycophenolate mofetil PO BID beginning on day 5 for 30 days.
  NK CELLS: Patients receive NK cells IV over 30 minutes on days 7 and 28.

SUMMARY:
This phase I/II study the side effects and efficacy of natural killer cells after donor stem cell transplant and how they treat patients with myeloid malignancies or lymphoproliferative disorders. Investigators expanded NK cells ex vivo with a non-feeder cell regimen to avoid the risk of infusion of feeder cells with expanded NK cells. Investigators infuse NK cells after myeloablative conditioning therapy. These cells may help decrease relapse of malignant disease, severe graft versus host disease, reactivation of certain viruses, and, therefore, prolong the survival of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with no matched related donor who has a related haploidentical donor identified (=< 7/8 allele match at the A, B, C, DR loci) who is willing to undergo a bone marrow harvest and an NK cell collection approximately 2 weeks of the recipient's admission for transplant; the donor must be 16 years of age or older and weigh at least 50kg.
2. Patients with one of the following diseases: acute myeloid leukemia (AML): a. first complete remission with high-risk features defined as (i) greater than 1 cycle of induction therapy required to achieve remission; (ii) preceding myelodysplastic syndrome (MDS); (iii) presence of FLT3 mutations or internal tandem duplication or other mutations associated with poor-risk AML (e.g., DNMT3A, TET2); (iv) French-American-British Classification (FAB) M6 or M7 classification; (v) adverse cytogenetics: -5, deletion (del) 5q, -7, del7q, abnormalities involving 3q, 9q, 11q, 20q, 21q, 17, +8 or complex karyotype (> 3 abnormalities); (vi) treatment-related AML, or b. second or more significant remission; patients beyond the second remission have to be in complete remission (CR) at transplant to be eligible, or c. primary induction failure with partial response to therapy who achieve adequate cytoreduction
3. Patients with myelodysplastic syndromes (MDS): a. de novo MDS with intermediate or high-risk International Prognostic Scoring System (IPSS) scores; patients with intermediate-1 features should have failed to respond to hypomethylating agent therapy or b. patients with treatment-related MDS
4. Chronic myeloid leukemia (CML): a. failed to achieve cytogenetic remission or have a cytogenetic relapse after treatment with at least 2 tyrosine kinase inhibitors, or b. accelerated phase or blast phase at any time
5. Lymphoma: a. refractory to or released from 1st line therapy, salvaged by 2nd line therapy, or b. high-risk lymphoma with CR to 1st line therapy.
6. Performance score of at least 70% by Karnofsky or 0 to 1 by Eastern Cooperative Oncology Group (ECOG) (age >= 12 years), or Lansky Play-performance scale of at least 70% or greater (age < 12 years)
7. Serum creatinine clearance equal to or more than 50 ml/min (calculated with Cockcroft-Gault formula)
8. Bilirubin equal or less than 1.5 mg/dl except for Gilbert's disease Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal to or less than 200 IU/ml for adults
9. Conjugated (direct) bilirubin less than 2 x upper limit of normal
10. Left ventricular ejection fraction equal to or greater than 40%
11. Diffusing capacity of the lung for carbon monoxide (DLCO) equal or greater than 50% predicted corrected for hemoglobin; for children =< 7 years of age who are unable to perform pulmonary function tests (PFT), oxygen saturation >= 92% on room air by pulse oximetry

11. Patient or patient's legal representative, parent(s), or guardian should provide written informed consent; the permission of a minor if participant's age is at least seven and less than eighteen years

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) positive; active hepatitis B or C
2. Uncontrolled infections; principal investigator (PI) is the final arbiter of this criterion Liver cirrhosis
3. Central nervous system (CNS) involvement within three months
4. Positive pregnancy test in a woman with childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization
5. Inability to comply with medical therapy or follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated doses (MTD) of natural killer (NK) cells | Up to day 70 post-transplant
  Primary Outcome Measures

SECONDARY OUTCOMES:
100-day treatment related mortality | Up to 100 days post-transplant
  Will be defined as death due to any cause without disease recurrence within 100 days post stem cell transplant (SCT). The method of Thall and Sung will be used, based on an historical rate of 35%.
Overall survival | Up to 2 years post-transplant
  Will be estimated using the Kaplan-Meier method, and distributions will be compared using log-rank tests.
Relapse-free survival | Up to 2 years post-transplant
  Will be estimated using the Kaplan-Meier method, and distributions will be compared using log-rank tests.
Time to engraftment | Up to 2 years post-transplant
  Will be estimated using the Kaplan-Meier method, and distributions will be compared using log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ji, MD, Principal Investigator — West China Hospital, Sichuan Uiversity
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China